CLINICAL TRIAL: NCT05998226
Title: Evaluation of a Virtual Antimicrobial Stewardship Team (VAT) on Antibiotic Prescriptions From Clinicians in Nursing Homes: A Multicenter Randomised Controlled Trial
Brief Title: VAT-2: Evaluation of a Virtual Antimicrobial Stewardship Team (VAT) on Antibiotic Prescriptions in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health Service of Amsterdam (Other Government)
Collaborators: Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC) (Other)
Responsible Party: Principal Investigator, Maarten Schim van der Loeff, Professor, Public Health Service of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: W23_041 #23.064
Record Dates: First submitted 2023-08-01; First posted 2023-08-18 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a multi-center, two-arm, randomized controlled trial to evaluate a virtual antibiotic stewardship team (VAT) compared to standard care in Dutch NHs. After assessment of eligibility, the participants (clinicians) in the study are randomized (1:1) to the standard of care arm or to the intervention arm (weekly VAT meeting for 9 months). Randomization will be done stratified on the basis of function (group 1. elderly care physicians, group 2. physicians in training to become a specialist/ other physicians, group 3. nurse practitioners/ physician assistants).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard care (control group) (No Intervention): The clinicians from the control arm do not participate in VAT meetings. The antibiotic prescriptions prescribed by clinicians in the control group are extracted from the prescription system after the study period. Two researchers independently extract the data from patient files, including any culture results, and assess the antibiotic use based on the algorithm from the current guidelines that are used in NHs.
- Virtual Antimicrobial stewardship Team (VAT) (intervention group) (Experimental): The VAT consists at least of a medical microbiologist and a clinician from the NH. Depending on the NH organization concerned and cooperation agreements, a pharmacist will or will not be involved. They conduct weekly consultations during 9 months to evaluate the antibiotic prescriptions of the clinician based on algorithms from current guidelines in use in the NH. This is an evaluation of standard care .
  Interventions: Other: Virtual Antimicrobial stewardship Team (VAT)

INTERVENTIONS:
Other: Virtual Antimicrobial stewardship Team (VAT) — The VAT consists of at least a clinical microbiologist and a clinician from the NH. Ideally, a pharmacist will also attend. They conduct a weekly (digital) meeting for nine months to evaluate the antibiotic prescriptions of the clinician attending the VAT meeting, based on a standardized protocol according to the current national infection treatment guidelines.
  Arms: Virtual Antimicrobial stewardship Team (VAT) (intervention group)

SUMMARY:
The Virtual Antimicrobial stewardship Team (VAT) study aims to evaluate, in a randomized controlled trial (RCT), the effect of a weekly virtual antimicrobial stewardship (AMS) intervention on the appropriateness of prescribing antibiotics for nursing home (NH) residents with urinary tract infections (UTI), respiratory tract infections (RTI) or skin and soft tissue infections (SSTI) compared to standard care for NH residents in Dutch NHs in the provinces of North-Holland and Flevoland. The secondary aim is to identify barriers and facilitators to implement a stewardship intervention and subsequently develop an implementation guide.

DETAILED DESCRIPTION:
Rationale: Antimicrobial stewardship interventions have been extensively studied in hospital settings and have proven effective in reducing the number of infections with multidrug resistant micro-organisms and are also cost-effective. Therefore, AMS teams are mandatory in Dutch hospitals.

The effectiveness of an antimicrobial stewardship intervention is variable in previous studies. Also due to the perceived high workload and costs, AMS has hardly been implemented in Dutch NHs. In order to take the next step towards implementation of AMS in NHs, causality between AMS and reduction in inappropriate antibiotic prescriptions should be demonstrated. The investigators want to evaluate the process and value of the VAT approach to facilitate optimal implementation of VAT in other NHs.

Objective: To demonstrate the efficacy of weekly virtual antimicrobial stewardship team meetings in reducing inappropriate antibiotic prescriptions in Dutch NHs.

Study design: randomized, non-blinded, controlled, multicenter trial.

Study population: Clinicians working in NHs in the provinces North Holland and Flevoland.

Intervention: The VAT consists of at least a clinical microbiologist and a clinician from the NH. Ideally, a pharmacist will also attend. They conduct a weekly (digital) meeting for nine months to evaluate the antibiotic prescriptions of the clinician attending the VAT meeting, based on a standardized protocol according to the current national guidelines.

Main study parameters/endpoints: The primary outcome is the number of inappropriate antibiotic prescriptions, assessed based on an algorithm of the current clinical infection treatment guidelines, antimicrobial susceptibility test results, and clinical characteristics. Each antibiotic prescription is a record and for each record will be assessed whether the antibiotic prescription is appropriate or not. Secondary outcome measures are the incidence rate (IR) of antibiotic prescriptions and facilitators and barriers to VAT implementation.

ELIGIBILITY:
Inclusion Criteria of clinicians:

* Working in nursing homes in the North Holland-Flevoland region and being authorized to prescribe.
* Agreeing to being randomized to intervention or control group.
* Working in a nursing home that has a medication prescription system from which prescriptions can easily be obtained for VAT meetings.
* Working in a nursing home that is connected to a microbiology lab, .that participates in this study and offers VAT meetings.
* Expected to be employed for at least four months from date of randomization.

Inclusion Criteria of antibiotic prescriptions:

• All prescriptions for antibiotics with a therapeutic indication regarding urinary tract infections, respiratory tract infections or skin and soft tissue infections for residents of nursing homes, prescribed by clinicians participating in the study, during the study period.

Exclusion Criteria of antibiotic prescriptions:

* Prescriptions for antibiotics with a prophylactic purpose.
* Prescriptions given by clinicians not participating in the study
* Prescriptions prescribed outside the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Inappropriate antibiotic prescriptions | 9 months
  The proportion of inappropriate antibiotic prescriptions in the intervention group compared to the control group (standard of care) according to the current guidelines algorithm.

SECONDARY OUTCOMES:
Incidence rate (IR) | 9 months
  Incidence rate (IR) of antibiotic prescriptions in each group.
Barriers and facilitators | 9 months
  Identify the barriers and facilitators for VAT implementation through questionnaires.
Barriers and facilitators | 9 months
  Identify the barriers and facilitators for VAT implementation through and in-depth interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Maarten MF Schim van der Loeff, Prof. dr., Principal Investigator — Public Health Service of Amsterdam
Locations (1):
- Public Health Service of Amsterdam, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paap KC, Kolodziej LM, van Buul LW, de Jong MD, van der Loeff MFS, Kuil SD. The impact of a weekly antimicrobial stewardship team intervention on antibiotic prescriptions in Dutch nursing homes: a protocol for a randomised controlled trial. Trials. 2025 Dec 29;26(1):587. doi: 10.1186/s13063-025-09303-w. PMID 41462319